CLINICAL TRIAL: NCT01656993
Title: Antiplatelet Activity of Aspirin in Infants After Aortopulmonary and Cavopulmonary Shunts
Status: Completed | Type: Observational
Sponsor: University of Utah (Other)
Responsible Party: Principal Investigator, Dongngan Truong, Pediatric Cardiology Fellow, University of Utah
Other Study IDs: 55107
Record Dates: First submitted 2012-07-26; First posted 2012-08-03 (Estimated); Last update posted 2017-05-05 (Actual); Status verified 2017-05

CONDITIONS: Congenital Heart Disease
Keywords: Aspirin; ASA; aortopulmonary shunt; cavopulmonary shunt; shunt; TEG; Antiplatelet
MeSH Terms: conditions — Heart Defects, Congenital

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- ASA activity: Participants (age 2.0 days to 12 months) undergoing cardiac surgery for a shunt and planned treatment with aspirin

SUMMARY:
Background: Blood clots cause poor outcomes, including death, in babies with heart defects that require a surgical connection ("shunt") to provide blood flow to their lungs. Aspirin (ASA) blocks the part of the blood that helps clots form (platelets). Aspirin is used in babies with shunts to prevent blood clots. The dose of aspirin given to babies is based on adult research. Because babies are different from adults, the investigators do not know if the dose is enough to block platelets, or if it is too much and may cause bleeding. The investigators can test the platelets using a blood test called Thromboelastography with Platelet Mapping (TEG-PM). This test needs a small amount of blood so it can be used in babies.

Hypothesis and Specific Aims: The investigators suspect the aspirin doses typically given babies are not enough to block platelets and prevent blood clots in their shunts. The investigators want to determine the percentage of babies whose platelets are not blocked enough (< 70% inhibition), by using TEG-PM. The investigators also want to determine how often bleeding or clots occur in babies receiving aspirin.

DETAILED DESCRIPTION:
Background: Aortopulmonary and cavopulmonary shunts ("shunts") are surgically placed to provide pulmonary blood flow in infants with congenital heart disease who require the shunt for survival. Thrombosis occurs in about 17% of these shunted infants (Li et al, 2007; Monagle et al, 2012) with an associated morbidity of 23% and mortality of 7%.(Li et al, 2007) One study reported a third of all deaths were from shunt thrombosis.(Fenton, 2003) Despite insufficient evidence to guide appropriate dosing, current thromboprophylaxis guidelines recommend aspirin (ASA) for thrombus prevention in these high-risk infants. No therapeutic monitoring exists to ensure consistent and effective anticoagulation and prevent over-anticoagulation to minimize bleeding complications. Previous studies examining the effectiveness of ASA in shunt thrombosis prevention have conflicting results. The most recent large, prospective observational study showed a significant association between ASA use and lower risk of thrombosis and death (Li et al, 2007), but the study was limited by lack of standardized ASA dosing and failure to include adverse events. To further complicate the picture, adult studies have described a phenomenon termed "ASA resistance," where thrombosis occurs despite ASA therapy.(Frelinger et al, 2008; Heistein et al, 2008; Szczeklik et al, 2005; Frelinger et al, 2006) ASA resistance has not been adequately studied in the pediatric population leading to a knowledge gap between therapeutic dosing and the adequate prevention of thrombosis combined with minimization of bleeding complications. Thromboelastography with Platelet Mapping (TEG-PM) is a blood test that specifically evaluates the percentage of inhibition of the arachidonic acid pathway targeted by ASA. It can be used for serial monitoring of the adequacy of anticoagulation with ASA in shunted infants and to provide evidence of safe and effective dosages for its use in other pediatric populations.

Hypothesis and Specific Aims:

Hypothesis: The investigators hypothesize that ASA dosing by current guidelines (1-5 mg/kg/day) favors protection from bleeding complications and fails to achieve adequate inhibition of the arachidonic acid pathway to prevent thrombosis.

Specific Aim 1: The primary aim is to determine the percentage of infants treated with ASA after shunt surgery who have adequate (> 70%) inhibition of the arachidonic acid pathway as measured by TEG-PM.

Outcome: The percentage of arachidonic inhibition, as measured by TEG-PM, at 3 designated time points after starting ASA postoperatively. Therefore, TEG-PM will be measured at these designated time points:

1. After the third dose of ASA
2. At the first post-operative cardiology clinic visit (between 2 and 4 weeks after hospital discharge)
3. At a follow-up cardiology clinic visit 3-6 months after the initiation of ASA

Specific Aim 2: The secondary aim is to describe the frequency of bleeding and thrombotic events while on ASA.

Outcome: The number of bleeding and thrombotic events from initiation of ASA therapy to end of study will be documented.

ASA administration: ASA will be initiated by the cardiac intensive care unit attending physician postoperatively, at a dose of 1-5 mg/kg/day, but no less than 20 mg per day; the initiation of ASA at 1-5 mg/kg/day is standard of care and recommended by the College of Chest Physicians (Monagle et al, 2012), albeit with limited evidence for its use. TEG-PM results obtained for research purposes will be available only to the research team. The dose of ASA will not be adjusted by results from the research TEG-PM. However, if bleeding or thrombosis occurs, TEG-PM is obtained by local practice and ASA dosing adjusted by the treating physician. If the dose of ASA is changed while the patient is hospitalized, TEG-PM will be obtained 2 hours after the third (adjusted or restarted) dose.

ELIGIBILITY:
Inclusion Criteria:

* Undergoing cardiac surgery for a shunt and planned treatment with aspirin
* Age 2.0 days to 12 months
* Consent of parent or guardian

Exclusion Criteria:

* Known or suspected congenital or acquired coagulation disorders (such as hemophilia, von Willebrands disease, Glansmans thrombasthenia).
* History of aspirin use within 7 days of surgery.
* Platelet count < 50K prior to surgery.
* Weight < 2.5 kg.
* Prematurity defined as gestational age < 37 weeks.

Ages: 2 Days to 12 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Infants undergoing cardiac surgery involving aortopulmonary and/or cavopulmonary shunts with planned aspirin treatment
Sampling Method: Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2012-11 (Actual); Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
The percentage of arachidonic acid inhibition of platelets, as measured by TEG-PM after the initiation of ASA. | TEG-PM will be measured after the third dose of ASA is given postoperatively. (up to 6 months after surgery)

SECONDARY OUTCOMES:
The percentage of arachidonic acid inhibition of platelets, as measured by TEG-PM at the first postoperative cardiology clinic visit. | The percentage of arachidonic acid inhibition will be measured at the first post-operative cardiology clinic vist (typically 2-4 weeks after hospital discharge)
The percentage of arachidonic acid inhibition of platelets, as measured by TEG-PM 3-6 months after surgery. | TEG-PM will be measured 3-6 months postoperatively to determine the percentage of arachidonic acid inhibition.
The number of bleeding and thrombotic events while patients are on ASA. | Patients will be monitored for bleeding and thrombotic events while on ASA for the duration of this study, thus for up to 1.5 years.

CONTACTS AND LOCATIONS:
Overall Officials: Dongngan Truong, MD, Principal Investigator — University of Utah / Primary Children's Medical Center
Locations (1):
- Primary Children's Medical Center, Salt Lake City, Utah, United States

REFERENCES:
- [Background] Li JS, Yow E, Berezny KY, Rhodes JF, Bokesch PM, Charpie JR, Forbus GA, Mahony L, Boshkov L, Lambert V, Bonnet D, Michel-Behnke I, Graham TP, Takahashi M, Jaggers J, Califf RM, Rakhit A, Fontecave S, Sanders SP. Clinical outcomes of palliative surgery including a systemic-to-pulmonary artery shunt in infants with cyanotic congenital heart disease: does aspirin make a difference? Circulation. 2007 Jul 17;116(3):293-7. doi: 10.1161/CIRCULATIONAHA.106.652172. Epub 2007 Jun 25. PMID 17592082
- [Background] Monagle P, Chan AKC, Goldenberg NA, Ichord RN, Journeycake JM, Nowak-Gottl U, Vesely SK. Antithrombotic therapy in neonates and children: Antithrombotic Therapy and Prevention of Thrombosis, 9th ed: American College of Chest Physicians Evidence-Based Clinical Practice Guidelines. Chest. 2012 Feb;141(2 Suppl):e737S-e801S. doi: 10.1378/chest.11-2308. PMID 22315277
- [Background] Fenton KN, Siewers RD, Rebovich B, Pigula FA. Interim mortality in infants with systemic-to-pulmonary artery shunts. Ann Thorac Surg. 2003 Jul;76(1):152-6; discussion 156-7. doi: 10.1016/s0003-4975(03)00168-1. PMID 12842531
- [Background] Frelinger AL, Li Y, Linden MD, Tarnow I, Barnard MR, Fox ML, Michelson AD. Aspirin 'resistance': role of pre-existent platelet reactivity and correlation between tests. J Thromb Haemost. 2008 Dec;6(12):2035-44. doi: 10.1111/j.1538-7836.2008.03184.x. Epub 2008 Oct 7. PMID 18983514
- [Background] Heistein LC, Scott WA, Zellers TM, Fixler DE, Ramaciotti C, Journeycake JM, Lemler MS. Aspirin resistance in children with heart disease at risk for thromboembolism: prevalence and possible mechanisms. Pediatr Cardiol. 2008 Mar;29(2):285-91. doi: 10.1007/s00246-007-9098-7. Epub 2007 Sep 25. PMID 17896127
- [Background] Szczeklik A, Musial J, Undas A, Sanak M, Nizankowski R. Aspirin resistance. Pharmacol Rep. 2005;57 Suppl:33-41. PMID 16415485
- [Background] Frelinger AL 3rd, Furman MI, Linden MD, Li Y, Fox ML, Barnard MR, Michelson AD. Residual arachidonic acid-induced platelet activation via an adenosine diphosphate-dependent but cyclooxygenase-1- and cyclooxygenase-2-independent pathway: a 700-patient study of aspirin resistance. Circulation. 2006 Jun 27;113(25):2888-96. doi: 10.1161/CIRCULATIONAHA.105.596627. Epub 2006 Jun 19. PMID 16785341